CLINICAL TRIAL: NCT07247747
Title: Turkish Validity and Reliability of Virtual Reality System Usability Questionnaire
Brief Title: Turkish Validity and Reliability of VRSUQ
Status: Not yet recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, enes tayyip benli, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-BENLI-007
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Virtual reality group: They will experience some virtual reality applications and carry out questionnaires to test the validity and reliability of the scale

SUMMARY:
The aim of this study is to conduct a Turkish validity and reliability study of the Virtual Reality System Usability Questionnaire (VRSUQ), which can evaluate virtual reality from various aspects by taking into account the characteristics of virtual reality and usability evaluation indicators.

DETAILED DESCRIPTION:
Virtual reality-based rehabilitation approaches are attracting increasing attention and research. It is a necessity and a challenge for researchers to demonstrate the degree of usability of existing or newly designed applications suitable for rehabilitation purposes. For this purpose, the System Usability Scale designed to evaluate the usability of simulations is used, but it does not contain items specifically for immersive virtual reality. The usability scale developed specifically for immersive virtual reality aims to fill this gap. This study was planned to conduct a Turkish validity and reliability study of this questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in the research
* To be between the ages of 18-50
* Ability to stand and walk independently

Exclusion Criteria:

* Scores below 24 on the mini mental test
* Scoring 10 and above on the simulator disease questionnaire
* People with amblyopia, strabismus and pathologies that interfere with focusing, depth perception or normal 3D vision
* Failure of the fly test in the Titmus test

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Bolu Abant Izzet Baysal University Faculty of Health Sciences will be held with the participation of students and academicians
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Virtual Reality System Usability Questionnaire | From enrollment to the second assesment at 2 weeks
  The Virtual Reality System Usability Questionnaire consists of usability evaluation indicators that reflect the characteristics of VR applications and the questionnaire consists of nine items. The Virtual Reality System Usability Questionnaire includes questions about the response time of the system, clarity of feedback and ease of error correction specific to VR systems. 9 items scored on a five-point Likert scale (1 = strongly disagree, 5 = strongly agree). Negative-worded items are reverse-coded. Final scores are converted to a 0-100 scale, with higher scores indicating better perceived usability.